CLINICAL TRIAL: NCT00575731
Title: Behavioral Strategies for Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Michaela Kiernan, Senior Research Scientist, Stanford University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: SU-11082007-857
Record Dates: First submitted 2007-12-16; First posted 2007-12-18 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Fine-Tuning (Experimental): 2-month intervention (8 lifestyle counseling classes)
  Interventions: Behavioral: Weight management strategies
- Record-Keeping (Active Comparator): 2-month intervention (8 lifestyle counseling classes)
  Interventions: Behavioral: Weight management strategies

INTERVENTIONS:
Behavioral: Weight management strategies

SUMMARY:
Although studies demonstrate that people who consistently keep detailed food records are more likely to maintain their weight, few people continue to keep records given the vigilant attention needed. This study will test the efficacy of an alternative approach to record keeping that may be easier for people to sustain and lead to better long-term weight management. We propose that obese adults who attempt to keep their weight within a clearly defined and personalized 'range', e.g., a 5-lb range between 200-205 pounds, will be more likely to continue weighing themselves and remain weight stable because they have learned to self-regulate, i.e., accurately monitor changes in their weight, alert themselves when they've gained too much weight, and 'finetune' their eating and physical activity in response, but with the minimum effort and attention necessary. The primary aim for this randomized trial will examine whether participants in an 8-week 'Fine-Tuning' program are more likely to weigh themselves over the 6-month study than participants in an 8-week traditional 'Record-Keeping' program.

DETAILED DESCRIPTION:
Although studies demonstrate that people who consistently keep detailed food records are more likely to maintain their weight, few people continue to keep records given the vigilant attention needed. This study will test the efficacy of an alternative approach to record keeping that may be easier for people to sustain and lead to better long-term weight management. We propose that obese adults who attempt to keep their weight within a clearly defined and personalized 'range', e.g., a 5-lb range between 200-205 pounds, will be more likely to continue weighing themselves and remain weight stable because they have learned to self-regulate, i.e., accurately monitor changes in their weight, alert themselves when they've gained too much weight, and 'finetune' their eating and physical activity in response, but with the minimum effort and attention necessary. The primary aim for this randomized trial will examine whether participants in an 8-week 'Fine-Tuning' program are more likely to weigh themselves over the 6-month study than participants in an 8-week traditional 'Record-Keeping' program.

ELIGIBILITY:
Inclusion Criteria:(a)Web screen: Men or women of any ethnic background; age 18 years or older; body mass index (BMI) 25-39; planning to remain in the area for the next six months; not pregnant or not planning to become pregnant within the next six months; has no history of heart disease, including stroke, heart attack, coronary artery bypass surgery, or balloon angioplasty; not currently under medical care for any of the following conditions: cardiovascular problems (stroke, heart attack, chest pain, bypass surgery, etc.); cancer (except skin cancer); diabetes; respiratory problems (chronic asthma, bronchitis, etc.); or psychiatric condition; not currently taking or stable on medications for vascular problems (such as high blood pressure); able to participate in physical activity; does not meet Diagnostic and Statistical Manual criteria for binge eating; does not have a health condition that requires a special diet; not participating in a weight-loss program; not participating in support groups that focus on weight and eating habits; not taking weight-loss medication; not participating in any other research trial; and willing to be randomly assigned to either intervention.

(b)Pre-randomization: Completes all of the following in a timely and thorough manner: baseline clinic visit, baseline questionnaires on the study website, and obtains medical approval for participation (if applicable). Exclusion Criteria:(a)Web screen: Men or women of any ethnic background; age 18 years or older; body mass index (BMI) 25-39; planning to remain in the area for the next six months; not pregnant or not planning to become pregnant within the next six months; has no history of heart disease, including stroke, heart attack, coronary artery bypass surgery, or balloon angioplasty; not currently under medical care for any of the following conditions: cardiovascular problems (stroke, heart attack, chest pain, bypass surgery, etc.); cancer (except skin cancer); diabetes; respiratory problems (chronic asthma, bronchitis, etc.); or psychiatric condition; not currently taking or stable on medications for vascular problems (such as high blood pressure); able to participate in physical activity; does not meet Diagnostic and Statistical Manual criteria for binge eating; does not have a health condition that requires a special diet; not participating in a weight-loss program; not participating in support groups that focus on weight and eating habits; not taking weight-loss medication; not participating in any other research trial; and willing to be randomly assigned to either intervention.

(b)Pre-randomization: Completes all of the following in a timely and thorough manner: baseline clinic visit, baseline questionnaires on the study website, and obtains medical approval for participation (if applicable).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-07; Primary Completion 2008-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Weighing attitudes and behavior | 6 months
Weight fluctuations | 6 months

SECONDARY OUTCOMES:
Psychological outcomes | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Kiernan, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States